CLINICAL TRIAL: NCT03059108
Title: Evaluation of B+ Surface on Early Loading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Pablo Galindo-Moreno, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 216CEIH2016
Record Dates: First submitted 2017-02-12; First posted 2017-02-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially | interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Loading (Experimental): Implant early loading: prosthesis delivery 4 weeks after implant placement
  Interventions: Procedure: Early Loading
- Conventional Loading (Active Comparator): Implant conventional loading: prosthesis delivery 8 weeks after implant placement
  Interventions: Procedure: Conventional Loading

INTERVENTIONS:
Procedure: Early Loading — The procedure in this group will consist on placing implant-supported restorations over the implants placed 4 weeks earlier. The device (dental implant) is of the same type in both groups.
  Arms: Early Loading
Procedure: Conventional Loading — The procedure in this group will consist on placing implant-supported restorations over the implants placed 8 weeks earlier. The device (dental implant) is of the same type in both groups.
  Arms: Conventional Loading

SUMMARY:
The trial is designed as a consecutive enrollment prospective one-center study. A minimum of 30 patients will be included in the study. At implant installation, the implant will be randomized to one of the groups (Control: conventional loading, 8 weeks; Test: early loading, 4 weeks). Samples of peri-implant crevicular fluid (PICF) and intrasulcular plaque will be collected at -14, 0 (Baseline: prosthesis delivery), 7 days and 1, 3, 6, 12 months. Prosthesis will be fabricated and delivered as usual, i.e., approximately two weeks after the impressions are taken.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 and ≤75 years old
* One missing tooth in the premolar or molar area with both opposing and adjacent teeth (mesial and distal).

Exclusion Criteria:

* One-stage bone augmentation
* Heavy smokers (>10 cigarettes/day)
* Uncontrolled type 1 or 2 diabetes (HgA1c>8)
* Known auto-immune or inflammatory disease
* Severe hematologic disorders, such as hemophilia or leukemia
* Local or systemic infection that may compromise normal healing (e.g., extensive periapical pathology)
* Liver or kidney dysfunction/failure
* Currently receiving cancer treatment or within 18 months from completion of radio- or chemotherapy
* Long-term history of oral bisphosphonates use (i.e., 10 years or more)
* History of intravenous bisphosphonates
* Long-term (>3 months) history of antibiotics or drugs known to alter the inflammation and/or immunological system
* Severe osseous diseases (e.g., Paget disease of bone)
* Pregnant women or nursing mothers
* Not able or not willing to follow instructions related to the study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Clinical success of B+-treated dental implants after conventional or early loading protocol as described by the International Congress of Oral Implantologists, Pisa Consensus Conference, 2007 | 12 months

SECONDARY OUTCOMES:
Change in marginal bone level around B+-treated implants after conventional or early loading protocol | 0 (Baseline: prosthesis delivery), 3, 6, and 12 months
Change in inflammatory markers in peri-implant crevicular fluid around B+-treated implants after conventional or early loading protocol | -14, 0 (Baseline: prosthesis delivery), 7 days and 1, 3, 6, 12 months
Change in the microbiological profile around B+-treated implants after conventional or early loading protocol | -14 (before impressions), 0 (Baseline: prosthesis delivery), 7 days and 1, 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Galindo-Moreno, DDS, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Facultad de Odontología, Granada, Spain

REFERENCES:
- [Result] Galindo-Moreno P, Gutierrez-Garrido L, Lopez-Chaichio L, Guerra-Lorenzo C, Rodriguez-Alvarez R, Padial-Molina M. Crestal bone changes around early vs. conventionally loaded implants with a multi-phosphonate coated surface: A randomized pilot clinical trial. Clin Oral Implants Res. 2021 Jan;32(1):75-87. doi: 10.1111/clr.13681. Epub 2020 Dec 18. PMID 33210771
- [Derived] Galindo-Moreno P, Gutierrez-Garrido L, Duarte J, Robles-Vera I, Martin-Morales N, O'Valle F, Olaechea A, Carrillo-Galvez AB, Padial-Molina M. Evolution in the Peri-Implant Oral Microbiome and Their Relationship to Long-Term Marginal Bone Loss: A Randomized Clinical Study. Clin Oral Implants Res. 2025 Jul;36(7):802-820. doi: 10.1111/clr.14426. Epub 2025 Mar 10. PMID 40062725